CLINICAL TRIAL: NCT03931343
Title: Randomized, Double Blind Trial of Thoracolumbar Interfascial Plane Block and Erector Spinae Plane Block for Adult Spinal Surgery
Brief Title: Comparison of Thoracolumbar Interfascial and Erector Spinae Plane Block on Analgesic Efficiency of After Spinal Surgery
Acronym: TALIPES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Yeşiltaş, İnstructor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S002
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Opioid Use
Keywords: Thoracolumbar interfascial block, Erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracolumbar interfascial plane block (Experimental): Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between multifidus and longissimus muscle with USG guidance
  Interventions: Procedure: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between multifidus and longissimus muscle with USG guidance
- Erectro spinae plane block (Active Comparator): Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between the erector spinae muscles and transverse process with USG guidance
  Interventions: Procedure: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between the erector spinae muscles and transverse process with USG guidance

INTERVENTIONS:
Procedure: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between multifidus and longissimus muscle with USG guidance — Thoracolumbar interfascial plane block: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between multifidus and longissimus muscle with USG guidance
  Other Names: Thoracolumbar interfascial plane block
  Arms: Thoracolumbar interfascial plane block
Procedure: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between the erector spinae muscles and transverse process with USG guidance — Erector spinae plane block: Bilateral 20 ml 0.25 % Bupivacaine with 2mg preservative free dexametasone and 5mcg/ml epinephrine injected between the erector spinae muscles and transverse process with USG guidance
  Other Names: Erector spinae plane block
  Arms: Erectro spinae plane block

SUMMARY:
Spinal surgery is typically associated with severe postoperative pain. Although the number of spinal surgeries has increased day by day, postoperative pain management have been limited. The recently described thoracolumbar interfacial plane block (TLIPB) has been reported to provide effective postoperative analgesia in spinal surgery. In addition, the recently described erector spinae plane block (ESPB) is obtained by applying the local anesthetic drug between the fascia of the spina muscles and the transverse process of the vertebrae. Anatomical and radiological investigations in fresh cadavers suggest that the potential place of influence of ESPB is dorsal and ventral spinal nerve roots. A small number of publications showing the analgesic efficacy of ESP in spinal surgery have been reported in the literature. In this study, the investigators aimed to compare the analgesic efficacy of TLIPB and ESPB in spinal surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75 years
2. ASA 1-2-3
3. Patients scheduled for elective surgery

Exclusion Criteria:

1. Patients with previous neurological disease symptoms (TIA, syncope, dementia, etc.)
2. Allergy to drugs
3. Major cardiac disease
4. Renal failure
5. Psychiatric disease
6. Patients who refuse to participate in the study
7. Chronic back and lower back pain

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hour
  The total amount of morphine given by patient controlled analgesia in 48 hours will be recorded.

SECONDARY OUTCOMES:
Pain intensity score at rest | 48 hour
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at postoperative 1, 3, 6, 12, 24, 48 hour. he NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of patient pain. Each item is scored 0-10( 0:no pain 10: pain as bad as can be )
Pain intensity score at movement | 48 hour
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at postoperative 1, 3, 6, 12, 24, 48 hour. he NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of patient pain. Each item is scored 0-10( 0:no pain 10: pain as bad as can be )
Time to first rescue analgesia | 48 hour
  If VAS is greater than 3, 25 mg of meperidine will be administered.
Postoperative nausea and vomiting | 48 hour
  Changes in Numeric Rank Score will be recorded at postoperative 1, 3, 6, 12, 24, 48 hour. Numeric rank score 0-3(0: no nausea and vomiting; 1:have nausea, no vomiting; 2:once vomiting attack; 3: have two or more vomiting attacks)
Patient satisfaction score | 48 hour
  Will be scored between 1-5 (1- very bad 5-very good).

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Yeşiltaş, Principal Investigator — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: No